CLINICAL TRIAL: NCT01524562
Title: HIV-Accelerated Liver Disease in Uganda
Brief Title: HIV Accelerated Liver Disease in Uganda
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912037; 12-I-N037
Record Dates: First submitted 2012-02-01; First posted 2012-02-02 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Fibrosis
Keywords: Fibrosis; Cirrhosis; Africa; Schistosomiasis; Aflatoxin; Liver Disease
MeSH Terms: conditions — Fibrosis; Schistosomiasis; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (2):
- Rakai Community Cohort: HIV Patients
- Rakai HIV Care Program: HIV Patients

SUMMARY:
Background:

- Liver disease is a leading cause of death in people who have the human immunodeficiency virus (HIV). It especially affects those who have both HIV and hepatitis B or C viruses. Most research on HIV-related liver disease has been conducted in North America and Europe. However, HIV-related liver disease in Uganda and other African nations may involve other diseases that are not common in the West, and may not involve hepatitis B or C. Researchers want to study HIV-related liver disease in Uganda to learn more about the differences between Western and African trends of this disease.

Objectives:

- To study HIV-related liver disease in rural Uganda.

Eligibility:

* Individuals at least 18 years of age who were tested for possible liver disease. Some participants will have HIV infection; others will be uninfected.
* All participants will be from rural areas of Uganda.

Design:

* Participants will have at least two study visits.
* Participants will have a physical exam and medical history. They will complete a questionnaire about health and quality of life. Blood, urine, and stool samples will be collected. Participants will also have a liver scan to check for liver scarring, and an ultrasound to take images of the liver.
* Participants who may have liver disease will visit a local hospital for more tests. A liver biopsy will be performed to collect liver tissue samples.

DETAILED DESCRIPTION:
With improved survival following the introduction of highly active antiretroviral therapy (HAART), liver disease has become a leading cause of death among HIV-infected persons in Western cohorts, primarily affecting those co-infected with hepatitis B or C viruses (HBV, HCV). However, data are sparse on liver disease in HIV-infected populations from Uganda and other African nations, where the etiologies of liver disease are broader and include aflatoxin, schistosomiasis and other infectious and environmental agents. Our previous noninvasive study in rural, Rakai, Uganda indicates that the prevalence of significant liver fibrosis is high among HIV-infected individuals (17%) and is 50% higher than in HIV-uninfected persons, although the prevalence of viral hepatitis B co-infection is low (5%). The study presented here is a biopsy-based study that follows up on these results with the objectives of defining the etiology of liver disease and describing the mechanisms of HIV-accelerated liver fibrosis in this setting.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Adults aged 18 and older
  2. Persons who are able and willing to provide informed consent
  3. Persons who have a transient elastography score >=9.0 kPa or have other evidence of liver disease, and who are willing to undergo an ultrasound and liver biopsy

     i) Other evidence of liver disease: Persons with an LSM <9.0 kPa who demonstrate liver transaminases at least 2-times greater than the upper limit of normal; those with persistently abnormal liver

     transaminases over a period of three months during the year preceding enrollment; those who show abnormalities on their ultrasound; those with other laboratory tests indicating the possibility of liver disease; and/or those who have a clinical or medical indication for a liver biopsy.
  4. Persons who are willing to have tissue samples undergo genetic testing
  5. Persons who agree to have samples stored for the purpose of future research

EXCLUSION CRITERIA:

1. Women who are pregnant
2. Persons with a cardiac device (i.e., pacemaker)
3. Participants who are not able to follow study instructions
4. Safety laboratory data indicating possible excess risk of bleeding including platelets <75,000 and an INR>=1.5. These safety laboratory values will be ascertained by obtaining a Complete Blood Count (CBC) and a Prothrombin Time (PT).
5. Evidence of decompensated liver disease including ascites, or hepatic encephalopathy
6. Persons who have any condition deemed, by the investigators, to be a contraindication to study participation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 786 (Actual)
Dates: Start 2011-12-20 (Actual); Primary Completion 2015-05-12 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Defining the eriology of liver disease | 2 years
  Describe the etiologiges and compare the pathogenesis of liver fibrosis in HIV-infected and HIV-uninfected persons wirh evidence of liver disease in rural, Rakai Uganda.

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Reynolds, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), 9000 Rockville Pi, Bethesda, Maryland, United States

REFERENCES:
- [Background] Salmon-Ceron D, Lewden C, Morlat P, Bevilacqua S, Jougla E, Bonnet F, Heripret L, Costagliola D, May T, Chene G; Mortality 2000 study group. Liver disease as a major cause of death among HIV infected patients: role of hepatitis C and B viruses and alcohol. J Hepatol. 2005 Jun;42(6):799-805. doi: 10.1016/j.jhep.2005.01.022. PMID 15973779
- [Background] Soriano V, Martin-Carbonero L, Garcia-Samaniego J, Puoti M. Mortality due to chronic viral liver disease among patients infected with human immunodeficiency virus. Clin Infect Dis. 2001 Nov 15;33(10):1793-5. doi: 10.1086/323009. No abstract available. PMID 11641832
- [Background] Lewden C, Salmon D, Morlat P, Bevilacqua S, Jougla E, Bonnet F, Heripret L, Costagliola D, May T, Chene G; Mortality 2000 study group. Causes of death among human immunodeficiency virus (HIV)-infected adults in the era of potent antiretroviral therapy: emerging role of hepatitis and cancers, persistent role of AIDS. Int J Epidemiol. 2005 Feb;34(1):121-30. doi: 10.1093/ije/dyh307. Epub 2004 Nov 23. PMID 15561752